CLINICAL TRIAL: NCT02157714
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study of PRX002 Administered By Intravenous Infusion in Patients With Parkinson's Disease
Brief Title: Multiple Ascending Dose Study of PRX002 in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prothena Biosciences Limited (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRX002-CL002
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- PRX002 (Experimental): PRX002
  Interventions: Drug: PRX002
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PRX002
  Arms: PRX002
Other: Placebo
  Arms: Placebo

SUMMARY:
This multiple ascending dose study is to determine safety, tolerability, pharmacokinetics and immunogenicity of PRX002 in approximately 60 patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease, Hoehn and Yahr 1-3
* Body weight range of ≥ 45kg/99 lbs to ≤ 110 kg/242 lbs
* Female subjects must be surgically sterile or post-menopausal or if of child-bearing potential must use contraception
* Male subjects and their partners of childbearing potential must use contraception

Exclusion Criteria:

* Significant cardiac history
* Abnormal MRI
* Significant laboratory abnormalities

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as determined by number of subjects with adverse events | up to 6 months
Determination of pharmacokinetics parameters | up to 6 months
  maximum concentration (Cmax)
Determination of pharmacokinetics parameters | up to 6 months
  time of the maximum measured concentration (Tmax)
Determination of pharmacokinetics parameters | up to 6 months
  area under the concentration-time curve from time zero to the last quantifiable concentration time-point (AUClast)
Determination of pharmacokinetics parameters | up to 6 months
  area under the concentration-time curve from time zero extrapolated to infinity (AUCinf)
Determination of pharmacokinetics parameters | up to 6 months
  elimination rate constant
Determination of pharmacokinetics parameters | up to 6 months
  terminal elimination half life (t½)
Determination of pharmacokinetics parameters | up to 6 months
  clearance (CL)
Determination of pharmacokinetics parameters | up to 6 months
  apparent volume of distribution (Vd)
Determination of pharmacokinetics parameters | up to 6 months
  average concentration over a dosing interval (Cav)
Determination of pharmacokinetics parameters | up to 6 months
  area under the plasma concentration-time curve for a dosing interval (AUCtau)
Determination of pharmacokinetics parameters | up to 6 months
  minimum observed concentration (Cmin)

SECONDARY OUTCOMES:
Immunogenicity as determined by measurement of anti-PRX002 antibodies | up to 3 months
  Multiple clinical and exploratory biomarkers will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Jay Soto, Study Director — Clinical Trials Prothena Biosciences Inc
Locations (8):
- United States (8):
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - MD Clinical, Hallandale, Florida
  - Compass Research, LLC, Orlando, Florida
  - QUEST Research Institute, Bingham Farms, Michigan
  - Oregon Health and Science University, Department of Neurology, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Jankovic J, Goodman I, Safirstein B, Marmon TK, Schenk DB, Koller M, Zago W, Ness DK, Griffith SG, Grundman M, Soto J, Ostrowitzki S, Boess FG, Martin-Facklam M, Quinn JF, Isaacson SH, Omidvar O, Ellenbogen A, Kinney GG. Safety and Tolerability of Multiple Ascending Doses of PRX002/RG7935, an Anti-alpha-Synuclein Monoclonal Antibody, in Patients With Parkinson Disease: A Randomized Clinical Trial. JAMA Neurol. 2018 Oct 1;75(10):1206-1214. doi: 10.1001/jamaneurol.2018.1487. PMID 29913017
- [Derived] Schenk DB, Koller M, Ness DK, Griffith SG, Grundman M, Zago W, Soto J, Atiee G, Ostrowitzki S, Kinney GG. First-in-human assessment of PRX002, an anti-alpha-synuclein monoclonal antibody, in healthy volunteers. Mov Disord. 2017 Feb;32(2):211-218. doi: 10.1002/mds.26878. Epub 2016 Nov 25. PMID 27886407